CLINICAL TRIAL: NCT02840201
Title: Sub-Clinical Atrial Fibrillation Biomarker (SCAF-b): A Sub-study of Apixaban for the Reduction of Thrombo-Embolism in Patients With Device-Detected Sub-Clinical Atrial Fibrillation (ARTESiA)
Brief Title: Sub-Clinical Atrial Fibrillation Biomarker Study
Acronym: SCAF-b
Status: Active, not recruiting | Type: Observational
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Collaborators: Population Health Research Institute (Other); Genome Canada (Other); Bristol-Myers Squibb (Industry); Pfizer (Industry); Medtronic (Industry); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Peter Liu, Chief Scientific Officer and VP of Research, Ottawa Heart Institute Research Corporation
Other Study IDs: 20150023
Record Dates: First submitted 2016-07-11; First posted 2016-07-21 (Estimated); Last update posted 2024-02-02 (Actual); Status verified 2024-02

CONDITIONS: Subclinical Atrial Fibrillation
Keywords: biomarkers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples will be collected for biomarker evaluation.
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a sub-study of the ARTESiA study registered as NCT01938248. This study is designed to validate biomarkers in subclinical atrial fibrillation and to determine if the prospective biomarker will be informative of the potential efficacy of treatment.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the most common cardiac rhythm disorder worldwide, and is gaining in prevalence. Currently, the treatment for atrial fibrillation is concentrated on patients with existing atrial fibrillation, and the reduction in risks of complications of stroke with anticoagulation. Furthermore, mechanical interventions such as atrial ablation procedures are fraught with inconsistent results. The availability of serum based biomarkers that can predict the early onset of atrial fibrillation, and also the ability to prognosticate risk, may help in the identification of patients at risk for AF complications early. This would also allow the identification of the patient population most suitable for the evaluation of possible future intervention strategies to prevent the onset of atrial fibrillation, and alter its natural history and complications.

Currently the best biomarkers in predicting atrial fibrillation risk are in fact markers for heart failure - NTproBNP and high sensitivity troponin. These markers are independent from CHA2DS2-VASc score. While this is very helpful, these markers will not be able to distinguish these 2 conditions because heart failure and atrial fibrillation often co-exist. The investigator's Cardiovascular Biomarker Discovery and Translation team has been using deep proteomic analysis of both human tissues and reprogrammed human stem cells to identify novel candidate biomarkers. This has been very successfully applied to diastolic heart failure, and there are now several new markers for this condition that have been validated across 3 populations. The investigators have several potential candidates for atrial fibrillation, but validation in the appropriate cohort, particularly those at the earliest risks of atrial fibrillation, will be most important.

The ARTESiA study is an ideal study setting to perform the biomarker validation, as the parent trial will recruit patients with silent atrial fibrillation detected only by dual-chamber pacemakers, defibrillators or insertable cardiac monitors. This would constitute a potentially earlier stage atrial fibrillation patient cohort, with known subsequent risks in a prospective fashion. The prospective evaluation of approved medications of aspirin and apixaban will also be helpful to determine if the prospective biomarker will be informative of the potential efficacy of treatment, or be unchanged by the treatment modalities.

ELIGIBILITY:
Inclusion Criteria:

* Permanent pacemaker or defibrillator (with or without resynchronization) or insertable cardiac monitor
* At least one episode of device-detected SCAF ≥ 6 minutes in duration but no single episode > 24 hours in duration at any time prior to enrollment. Any atrial high rate episode with average > 175 beats/min will be considered as SCAF. No distinction will be made between atrial fibrillation and atrial flutter. SCAF requires electrogram confirmation (at least one episode) unless ≥ 6 hours in duration
* Age ≥ 55 years
* Risk Factor(s) for Stroke:

Previous stroke, TIA or systemic arterial embolism OR Age at least 75 OR Age 65-74 with at least 2 other risk factors OR Age 55-64 with at least 3 other risk factors

Other risk factors are:

* Hypertension
* CHF
* Diabetes
* Vascular disease (i.e. CAD, PAD or Aortic Plaque)
* Female
* Must be from a participating Canadian recruitment centre
* Consent to participate in the ARTESiA parent study

Exclusion Criteria:

* Clinical atrial fibrillation documented by surface ECG (12 lead ECG, Telemetry, Holter) lasting ≥ 6 minutes, with or without clinical symptoms
* Mechanical valve prosthesis, recent (within past 6 months) deep vein thrombosis or pulmonary embolism or other condition requiring treatment with an anticoagulant
* Allergy to aspirin or apixaban
* Severe renal insufficiency (serum creatinine > 2.5 mg/dL [221 μmol/L] or a calculated creatinine clearance < 25 ml/min)
* Serious bleeding in the last 6 months or at high risk of bleeding (this includes, but is not limited to: prior intracranial hemorrhage, active peptic ulcer disease, clinically significant thrombocytopenia or anemia, recent stroke within past 10 days, documented hemorrhagic tendencies or blood dyscrasias)
* Moderate to severe hepatic impairment
* Ongoing need for combination therapy with aspirin and clopidogrel (or other combination of two platelet inhibitors)
* Meets criteria for requiring lower dose of apixaban AND also has ongoing need for strong inhibitors of both CYP3A4 and P-glycoprotein (e.g., ketoconazole, itraconazole, ritonavir or clarithromycin)
* Ongoing need for strong inducers of both CYP3A4 and P-glycoprotein (e.g., rifampin, carbamazepine, phenytoin, St. John's wort)
* Received an investigational drug in the past 30 days
* Participants considered by the investigator to be unsuitable for the study for any of the following reasons:
* Not agreeable for treatment with either aspirin or apixaban or anticipated to have poor compliance on study drug treatment
* Unwilling to attend study follow-up visits
* Life expectancy less than 2 years due to concomitant disease
* Women who are pregnant, breast-feeding or of child-bearing potential without an acceptable form of contraception in place (sterilization, abstinence or other method with less than 1% failure rate)

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Canadian patients participating in the ARTESiA study will be recruited for this sub-study.
Sampling Method: Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2017-06-26 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
The burden of silent atrial fibrillation as recorded on implanted devices in patients | 3 years
  as predicted by levels of proBNP, hsTnT and additional novel marker candidates

SECONDARY OUTCOMES:
The time related onset of complications | 3 years
  complications include embolic stroke, cerebral hemorrhage, myocardial infarction, heart failure and cardiac death, as predicted by both novel and known biomarkers outlined above.

OTHER OUTCOMES:
Comparison of time related onset of complications between those receiving aspirin versus apixaban. | 3 years
  complications such as embolic stroke, cerebral hemorrhage, myocardial infarction, heart failure and cardiac death will be compared between participants taking aspirin versus those taking apixaban

CONTACTS AND LOCATIONS:
Overall Officials: Peter Liu, MD, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No